CLINICAL TRIAL: NCT02887183
Title: A 52 Week, Open Label Evaluation of the Effects of Sacubitril/Valsartan (LCZ696) Therapy on Biomarkers, Myocardial Remodeling and Patient-reported Outcomes in Heart Failure With Reduced Left Ventricular Ejection Fraction.
Brief Title: Effects of Sacubitril/Valsartan Therapy on Biomarkers, Myocardial Remodeling and Outcomes.
Acronym: PROVE-HF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CLCZ696BUS13
Record Dates: First submitted 2016-08-29; First posted 2016-09-02 (Estimated); Results first posted 2019-12-05 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-10

CONDITIONS: Heart Failure
Keywords: Heart failure; Reduced left ventricular ejection fraction; HFrEF; NT-proBNP; Cardiac remodeling; sacubitril/valsartan; KCCQ; biomarkers
MeSH Terms: conditions — Heart Failure | interventions — sacubitril and valsartan sodium hydrate drug combination; sacubitril; Valsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (1):
- LCZ696(sacubitril/valsartan) (Other): Subjects received sacubitril/valsartan (LCZ696) on Day 1. The initial dose was determined by the investigator and per the approved indication described in the United States prescribing information/package insert (USPI). The three doses available were: 24/26 mg (Dose Level 1), 49/51mg (Dose Level 2) and 97/103mg (Dose Level 3).
  Titration of the dosage were performed per USPI at 2 to 4 week intervals as clinically tolerated until maximal tolerated or target dosage was achieved. Target dosage was sacubitril/valsartan 97/103 mg twice daily.
  Interventions: Drug: LCZ696 (sacubitril/valsartan)

INTERVENTIONS:
Drug: LCZ696 (sacubitril/valsartan) — LCZ696 (sacubitril/valsartan) was supplied as unscored, ovaloid, film-coated oral tablets in the strengths of 24/26 mg, 49/51 mg, 97/103 mg to be taken twice daily (bid)

SUMMARY:
This study was to determine early and more chronic changes in concentrations of biomarkers related to mechanisms of action (MOA) and effects of sacubitril/valsartan therapy over a period of 12 months, and correlated these biomarker changes with cardiac remodeling parameters, patient-reported outcomes and cardiovascular outcomes.

ELIGIBILITY:
Inclusion Criteria:

Based on the USPI for sacubitril/valsartan, subjects eligible for inclusion in this study must fulfill all of the following criteria at screening and baseline:

1. Written informed consent must be obtained before any assessment is performed.
2. Men and women ≥ 18 years of age.
3. LVEF ≤ 40% subjects who are candidates for on-label sacubitril/valsartan treatment per standard of care.
4. New York Heart Association (NYHA) Functional class II-IV.
5. LVEF ≤40% via any local measurement within the past 6 months using echocardiography, multi gated acquisition scan (MUGA), CT scanning, MRI or ventricular angiography provided no subsequent study documenting an EF of >40%. If the EF measurement is expressed as a value range, the average of the range endpoint values should be used as the EF.
6. If a subject is on a loop diuretic, they must be on a stable dose for 2 weeks prior to baseline.

Key Exclusion Criteria:

Subjects fulfilling any of the following criteria, at screening and prior to dispensing of study drug, are not eligible for inclusion in this study. No additional exclusions may be applied by the investigator, in order to ensure that the study population will be representative of all eligible subjects/subjects.

1. pregnant or nursing women
2. women of child bearing potential not using highly effective method of contraception during dosing and for 7 days after stopping study medication
3. History of hypersensitivity to any of the study drugs, including history of hypersensitivity to drugs of similar chemical classes, or allergy to angiotensin converting enzyme inhibitor (ACEIs), Angiotensin II Receptor Blockers (ARBs), or Neutral endopeptidase (NEP) inhibitors as well as known or suspected contraindications to the study drugs.
4. History of angioedema drug related or otherwise.
5. Requirement of treatment with either ACE inhibitor and/or ARB.
6. Subjects with a heart transplant or ventricular assistance device (VAD) or intent to transplant (on transplant list) or implant a VAD.
7. Subjects with a cardio resynchronization therapy devices (CRT/CRT-D) implanted within 6 months of screening visit.
8. Subjects who are currently taking inotropic agents.
9. Current or prior treatment with sacubitril/valsartan.
10. Subjects taking medications prohibited by the protocol.
11. Subjects with diabetes mellitus who are taking aliskiren.
12. Use of other investigational drugs within 5 half-lives of enrollment, or within 30 days until the expected pharmacodynamic effect has returned to baseline, whichever is longer.
13. Concomitant use of nesiritide.
14. Bile acid sequestering agents such as cholestyramine or colestipol are prohibited to avoid interference with study drug absorption.
15. Any hospital admission/discharge related to heart failure within 2 weeks prior to baseline.
16. The use of outpatient or inpatient i.v. diuretic therapy within 2 weeks prior to baseline.
17. Enrollment in another clinical trial within 30 days of screening.
18. Potassium > 5.2 mEq/L at screening.
19. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within one year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 794 (Actual)
Dates: Start 2016-10-25 (Actual); Primary Completion 2018-10-22 (Actual); Study Completion 2018-10-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (69):
- United States (69):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Fort Payne, Alabama
  - Novartis Investigative Site, Guntersville, Alabama
  - Novartis Investigative Site, Bakersfield, California
  - Novartis Investigative Site, Long Beach, California
  - Novartis Investigative Site, Los Alamitos, California
  - Novartis Investigative Site, Sylmar, California
  - Novartis Investigative Site, West Haven, Connecticut
  - Novartis Investigative Site, Belle Glade, Florida
  - Novartis Investigative Site, Bradenton, Florida
  - Novartis Investigative Site, Hollywood, Florida
  - Novartis Investigative Site, Homestead, Florida
  - Novartis Investigative Site, Jupiter, Florida
  - Novartis Investigative Site, Lake Worth, Florida
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Port Orange, Florida
  - Novartis Investigative Site, Wellington, Florida
  - Novartis Investigative Site, Arlington Heights, Illinois
  - Novartis Investigative Site, Aurora, Illinois
  - Novartis Investigative Site, Lombard, Illinois
  - Novartis Investigative Site, Oak Lawn, Illinois
  - Novartis Investigative Site, Louisville, Kentucky
  - Novartis Investigative Site, Owensboro, Kentucky
  - Novartis Investigative Site, Crowley, Louisiana
  - Novartis Investigative Site, Shreveport, Louisiana
  - Novartis Investigative Site, West Monroe, Louisiana
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Columbia, Maryland
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Haverhill, Massachusetts
  - Novartis Investigative Site, Springfield, Massachusetts
  - Novartis Investigative Site, Kalamazoo, Michigan
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, Belzoni, Mississippi
  - Novartis Investigative Site, Jackson, Mississippi
  - Novartis Investigative Site, Southhaven, Mississippi
  - Novartis Investigative Site, Bozeman, Montana
  - Novartis Investigative Site, Lincoln, Nebraska
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Nashua, New Hampshire
  - Novartis Investigative Site, Buffalo, New York
  - Novartis Investigative Site, Lake Success, New York
  - Novartis Investigative Site, Potsdam, New York
  - Novartis Investigative Site, The Bronx, New York
  - Novartis Investigative Site, Greensboro, North Carolina
  - Novartis Investigative Site, Hickory, North Carolina
  - Novartis Investigative Site, Winston-Salem, North Carolina
  - Novartis Investigative Site, Hillsboro, Oregon
  - Novartis Investigative Site, Oregon City, Oregon
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Camp Hill, Pennsylvania
  - Novartis Investigative Site, Wyomissing, Pennsylvania
  - Novartis Investigative Site, Yardley, Pennsylvania
  - Novartis Investigative Site, Simpsonville, South Carolina
  - Novartis Investigative Site, Germantown, Tennessee
  - Novartis Investigative Site, Austin, Texas
  - Novartis Investigative Site, Beaumont, Texas
  - Novartis Investigative Site, Bryan, Texas
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Hunstville, Texas
  - Novartis Investigative Site, McKinney, Texas
  - Novartis Investigative Site, Sherman, Texas
  - Novartis Investigative Site, Tomball, Texas
  - Novartis Investigative Site, Tyler, Texas
  - Novartis Investigative Site, White River Junction, Vermont
  - Novartis Investigative Site, Midlothian, Virginia
  - Novartis Investigative Site, Richmond, Virginia
  - Novartis Investigative Site, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Myhre PL, Liu Y, Kulac IJ, Claggett BL, Prescott MF, Felker GM, Butler J, Pina IL, Rouleau JL, Zile MR, McMurray JJV, Ward JH, Solomon SD, Januzzi JL. Changes in mid-regional pro-adrenomedullin during treatment with sacubitril/valsartan. Eur J Heart Fail. 2023 Aug;25(8):1396-1405. doi: 10.1002/ejhf.2957. Epub 2023 Jul 11. PMID 37401523
- [Derived] Mohebi R, Liu Y, Felker GM, Prescott MF, Pina IL, Butler J, Ward JH, Solomon SD, Januzzi JL. Prediction of Left Ventricular Ejection Fraction Change Following Treatment With Sacubitril/Valsartan. JACC Heart Fail. 2023 Jan;11(1):44-54. doi: 10.1016/j.jchf.2022.09.009. Epub 2022 Nov 9. PMID 36599549
- [Derived] Murphy SP, Ward JH, Pina IL, Felker GM, Butler J, Maisel AS, Meng X, Prescott MF, Solomon SD, Januzzi JL. Age Differences in Effects of Sacubitril/Valsartan on Cardiac Remodeling, Biomarkers, and Health Status. JACC Heart Fail. 2022 Dec;10(12):976-988. doi: 10.1016/j.jchf.2022.07.001. Epub 2022 Sep 7. PMID 36456072
- [Derived] Mohebi R, Liu Y, Pina IL, Prescott MF, Butler J, Felker GM, Ward JH, Solomon SD, Januzzi JL Jr. Dose-Response to Sacubitril/Valsartan in Patients With Heart Failure and Reduced Ejection Fraction. J Am Coll Cardiol. 2022 Oct 18;80(16):1529-1541. doi: 10.1016/j.jacc.2022.08.737. PMID 36229089
- [Derived] Myhre PL, Prescott MF, Claggett B, Felker GM, Butler J, Pina IL, Maisel AS, Williamson KM, Ward JH, Solomon SD, Januzzi JL. Comparative Effect of Angiotensin Receptor Neprilysin Inhibition on B-type Natriuretic Peptide Levels Measured by Three Different Assays: The PROVE-HF Study. Clin Chem. 2022 Nov 3;68(11):1391-1398. doi: 10.1093/clinchem/hvac148. PMID 36103292
- [Derived] Myhre PL, Prescott MF, Murphy SP, Fang JC, Mitchell GF, Ward JH, Claggett B, Desai AS, Solomon SD, Januzzi JL. Early B-Type Natriuretic Peptide Change in HFrEF Patients Treated With Sacubitril/Valsartan: A Pooled Analysis of EVALUATE-HF and PROVE-HF. JACC Heart Fail. 2022 Feb;10(2):119-128. doi: 10.1016/j.jchf.2021.09.007. Epub 2022 Jan 12. PMID 35115085
- [Derived] Murphy SP, Prescott MF, Maisel AS, Butler J, Pina IL, Felker GM, Ward JH, Williamson KM, Camacho A, Kandanelly RR, Solomon SD, Januzzi JL. Association Between Angiotensin Receptor-Neprilysin Inhibition, Cardiovascular Biomarkers, and Cardiac Remodeling in Heart Failure With Reduced Ejection Fraction. Circ Heart Fail. 2021 Jun;14(6):e008410. doi: 10.1161/CIRCHEARTFAILURE.120.008410. Epub 2021 May 15. PMID 33998243
- [Derived] Khan MS, Felker GM, Pina IL, Camacho A, Bapat D, Ibrahim NE, Maisel AS, Prescott MF, Ward JH, Solomon SD, Januzzi JL, Butler J. Reverse Cardiac Remodeling Following Initiation of Sacubitril/Valsartan in Patients With Heart Failure With and Without Diabetes. JACC Heart Fail. 2021 Feb;9(2):137-145. doi: 10.1016/j.jchf.2020.09.014. Epub 2020 Dec 9. PMID 33309581
- [Derived] Murphy SP, Prescott MF, Camacho A, Iyer SR, Maisel AS, Felker GM, Butler J, Pina IL, Ibrahim NE, Abbas C, Burnett JC Jr, Solomon SD, Januzzi JL. Atrial Natriuretic Peptide and Treatment With Sacubitril/Valsartan in Heart Failure With Reduced Ejection Fraction. JACC Heart Fail. 2021 Feb;9(2):127-136. doi: 10.1016/j.jchf.2020.09.013. Epub 2020 Nov 11. PMID 33189632
- [Derived] Pina IL, Camacho A, Ibrahim NE, Felker GM, Butler J, Maisel AS, Prescott MF, Williamson KM, Claggett BL, Desai AS, Solomon SD, Januzzi JL; PROVE-HF Investigators. Improvement of Health Status Following Initiation of Sacubitril/Valsartan in Heart Failure and Reduced Ejection Fraction. JACC Heart Fail. 2021 Jan;9(1):42-51. doi: 10.1016/j.jchf.2020.09.012. Epub 2020 Nov 11. PMID 33189630
- [Derived] Ibrahim NE, Pina IL, Camacho A, Bapat D, Felker GM, Maisel AS, Butler J, Prescott MF, Abbas CA, Solomon SD, Januzzi JL Jr; Prospective Study of Biomarkers, Symptom Improvement and Ventricular Remodeling During Entresto Therapy for Heart Failure (PROVE-HF) Study Investigators. Racial and Ethnic Differences in Biomarkers, Health Status, and Cardiac Remodeling in Patients With Heart Failure With Reduced Ejection Fraction Treated With Sacubitril/Valsartan. Circ Heart Fail. 2020 Nov;13(11):e007829. doi: 10.1161/CIRCHEARTFAILURE.120.007829. Epub 2020 Oct 3. PMID 33016100
- [Derived] Januzzi JL Jr, Prescott MF, Butler J, Felker GM, Maisel AS, McCague K, Camacho A, Pina IL, Rocha RA, Shah AM, Williamson KM, Solomon SD; PROVE-HF Investigators. Association of Change in N-Terminal Pro-B-Type Natriuretic Peptide Following Initiation of Sacubitril-Valsartan Treatment With Cardiac Structure and Function in Patients With Heart Failure With Reduced Ejection Fraction. JAMA. 2019 Sep 17;322(11):1085-1095. doi: 10.1001/jama.2019.12821. PMID 31475295
- [Derived] Januzzi JL, Butler J, Fombu E, Maisel A, McCague K, Pina IL, Prescott MF, Riebman JB, Solomon S. Rationale and methods of the Prospective Study of Biomarkers, Symptom Improvement, and Ventricular Remodeling During Sacubitril/Valsartan Therapy for Heart Failure (PROVE-HF). Am Heart J. 2018 May;199:130-136. doi: 10.1016/j.ahj.2017.12.021. Epub 2018 Feb 13. PMID 29754651
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=511

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 1031 patients screened for the study, 795 completed screening and were enrolled. One (1) patient completed screening but withdrew consent and did not enter the treatment phase. Therefore, the Full Analysis Set and the Safety Set was based on 794 patients.
Period: Overall Study
Arm/Group | LCZ696(Sacubitril/Valsartan)
Started | 795
Full Analysis Set | 794
Completed | 654
Not Completed | 141
Not completed — Adverse Event | 44
Not completed — Death | 30
Not completed — Pregnancy | 1
Not completed — Protocol Violation | 6
Not completed — Technical Problems | 2
Not completed — Lost to Follow-up | 13
Not completed — Physician Decision | 10
Not completed — Withdrawal by Subject | 35

BASELINE CHARACTERISTICS:
Population: One (1) patient completed screening but withdrew consent and did not enter the treatment phase.
Arm/Group | LCZ696(Sacubitril/Valsartan)
Number analyzed (Participants) | 794
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 369
  >=65 years | 425
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 226
  Male | 568
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 180
  White | 581
  More than one race | 0
  Unknown or Not Reported | 27

OUTCOME MEASURES:

1. Primary Outcome: Change in Concentration of N-terminal Pro-brain Natriuretic Peptide (NT-proBNP) From Baseline to One Year
Description: Change in concentration of N-terminal pro-brain natriuretic peptide (NT-proBNP) from baseline to one year
Time Frame: Baseline, one year
Population: Full Analysis Set
Measure: Geometric Mean (Full Range); unit: pg/mL
Arm/Group | LCZ696(Sacubitril/Valsartan)
Number analyzed (Participants) | 794
pg/mL | 0.5905 [0.5470 to 0.6375]
Statistical Analysis 1: Comparison: LCZ696(Sacubitril/Valsartan); Test type: Other; p < .0001, ANCOVA; Least Squared Geometric Mean Ratio = 0.6320, 95% CI 2-sided [0.5865 to 0.6810]

2. Primary Outcome: Change in Left Atrial Volume Index (LAVi), Left Ventricular End Diastolic Volume Index (LVEDVi), Left Ventricular End Systolic Volume Index (LVESVi), and From Baseline to One Year
Description: Change in left atrial volume index (LAVi), left ventricular end diastolic volume index (LVEDVi), left ventricular end systolic volume index (LVESVi), and from baseline to one year
Time Frame: Baseline, one Year
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: mL/m^2
Arm/Group | LCZ696(Sacubitril/Valsartan)
Number analyzed (Participants) | 794
mL/m^2
  LAVi: number analyzed (Participants) | 613
  LAVi | -7.57 (6.06)
  LVEDVi: number analyzed (Participants) | 629
  LVEDVi | -12.33 (8.89)
  LVESVi: number analyzed (Participants) | 629
  LVESVi | -15.35 (9.61)
Statistical Analysis 1: Comparison: LCZ696(Sacubitril/Valsartan); LAVi; Test type: Other; p < .0001, ANCOVA; Least Squared Mean = -7.57, 95% CI 2-sided [-7.98 to -7.15]
Statistical Analysis 2: Comparison: LCZ696(Sacubitril/Valsartan); LVEDVi; Test type: Other; p < .0001, ANCOVA; Least Squared Mean = -12.25, 95% CI 2-sided [-12.92 to -11.58]
Statistical Analysis 3: Comparison: LCZ696(Sacubitril/Valsartan); LVESVi; Test type: Other; p < .0001, ANCOVA; Least Squared Mean = -15.29, 95% CI 2-sided [-16.03 to -14.55]

3. Primary Outcome: Change in Left Ventricular Ejection Fraction (LVEF) From Baseline to One Year
Description: Change in Left ventricular ejection fraction (LVEF) from baseline to one year. LVEF is a measurement expressed as a percentage of how much blood the left ventricle pumps out with each contraction.
Time Frame: Baseline, one year
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | LCZ696(Sacubitril/Valsartan)
Number analyzed (Participants) | 794
Percentage | 9.38 (6.85)
Statistical Analysis 1: Comparison: LCZ696(Sacubitril/Valsartan); Test type: Other; p < .001, ANCOVA; Least Squared Mean = 9.37, 95% CI 2-sided [8.84 to 9.90]

4. Primary Outcome: Change in Log-transformed NT-proBNP and Change in Structural Cardiac Measurements LVESVi, LVEDVi, LAVi, and LVEF From Baseline to One Year
Description: Pearson's correlation coefficient was calculated between change in log-transformed NT-proBNP and change in structural cardiac measurements LVESVi, LVEDVi, LAVi, and LVEF from baseline to one year.
Time Frame: Baseline, one year
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Pearson's Correlation
Arm/Group | LCZ696(Sacubitril/Valsartan)
Number analyzed (Participants) | 794
Pearson's Correlation
  LVESVi: number analyzed (Participants) | 595
  LVESVi | 0.405 [0.335 to 0.470]
  LVEDVi: number analyzed (Participants) | 595
  LVEDVi | 0.320 [0.246 to 0.391]
  LAVi: number analyzed (Participants) | 579
  LAVi | 0.263 [0.186 to 0.338]
  LVEF: number analyzed (Participants) | 596
  LVEF | -0.381 [-0.448 to -0.310]
Statistical Analysis 1: Comparison: LCZ696(Sacubitril/Valsartan); LVESVi, LVEDVi, LAVi. LVEF; Test type: Other — Pearson's Correlation; p < .0001, t-test, 2 sided

5. Secondary Outcome: Change in Log-transformed NT-proBNP Concentration and Change in Echocardiographic Measurements LVESVi, LVEDVi, LAVi, and LVEF From Baseline to Month 6
Description: Pearson's correlation coefficient was calculated between change in log-transformed NT-proBNP and change in echocardiographic measurements LVESVi, LVEDVi, LAVi, and LVEF from baseline to Month 6
Time Frame: Baseline, Month 6
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Pearson's Correlation
Arm/Group | LCZ696(Sacubitril/Valsartan)
Number analyzed (Participants) | 794
Pearson's Correlation
  LVESVi: number analyzed (Participants) | 650
  LVESVi | 0.233 [0.159 to 0.305]
  LVEDVi: number analyzed (Participants) | 650
  LVEDVi | 0.164 [0.088 to 0.238]
  LAVi: number analyzed (Participants) | 625
  LAVi | 0.190 [0.113 to 0.264]
  LVEF: number analyzed (Participants) | 651
  LVEF | -0.226 [-0.298 to -0.152]
Statistical Analysis 1: Comparison: LCZ696(Sacubitril/Valsartan); LVESVi, LVEDVi, LAVi. LVEF; Test type: Other — Pearson's Correlation; p < .0001, t-test, 2 sided

6. Secondary Outcome: Change From Baseline in Concentration of N-terminal Pro-brain Natriuretic Peptide (NT-proBNP) and Change in Change in Left Atrial Volume Index (LAVi) by Selected Groups of Interest at Month 6
Description: Pearson's correlation coefficient to examine the association between change in log-transformed NT-proBNP and LAVi from baseline to 6 months overall in subgroups of interest, these subgroups are:
  1. Subjects with HFrEF and "low" NT-proBNP (<600 if not hospitalized or <400 if hospitalized) or "low" BNP (<150 if not hospitalized, <100 if hospitalized) at baseline.
  2. Subjects with new onset HF and/or RAAS naïve.
  3. Subjects who are not receiving the target sacubitril/valsartan dose.
Time Frame: Baseline, Month 6
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Pearson's Correlation Coefficient
Arm/Group | LCZ696(Sacubitril/Valsartan)
Number analyzed (Participants) | 794
Pearson's Correlation Coefficient
  Subjects with new onset HF and/or RAAS naïve: number analyzed (Participants) | 90
  Subjects with new onset HF and/or RAAS naïve | 0.487 [0.311 to 0.631]
  Subjects with HFrEF and "low" NT-proBNP: number analyzed (Participants) | 239
  Subjects with HFrEF and "low" NT-proBNP | 0.228 [0.105 to 0.345]
  Subjects not receiving target dose: number analyzed (Participants) | 202
  Subjects not receiving target dose | 0.117 [-0.021 to 0.251]
Statistical Analysis 1: Comparison: LCZ696(Sacubitril/Valsartan); Subjects with new onset HF and/or RAAS naïve; Test type: Other — Pearson's Correlation; p < .0001, t-test, 2 sided
Statistical Analysis 2: Comparison: LCZ696(Sacubitril/Valsartan); Subjects with HFrEF and "low" NT-proBNP; Test type: Other — Pearson's Correlation; p = 0.0003, t-test, 2 sided
Statistical Analysis 3: Comparison: LCZ696(Sacubitril/Valsartan); Subjects not receiving target dose; Test type: Other — Pearson's Correlation; p = 0.0956, t-test, 2 sided

7. Secondary Outcome: Change From Baseline in Concentration of N-terminal Pro-brain Natriuretic Peptide (NT-proBNP) and Change in Left Ventricular End Systolic Volume Index (LVESVi) by Selected Groups of Interest at Month 6
Description: Pearson's correlation coefficient to examine the association between change in log-transformed NT-proBNP and LVESVi from baseline to 6 months overall in subgroups of interest, these subgroups are:
  1. Subjects with HFrEF and "low" NT-proBNP (<600 if not hospitalized or <400 if hospitalized) or "low" BNP (<150 if not hospitalized, <100 if hospitalized) at baseline.
  2. Subjects with new onset HF and/or RAAS naïve.
  3. Subjects who are not receiving the target sacubitril/valsartan dose.
Time Frame: Baseline, Month 6
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Pearson's Correlation Coefficient
Arm/Group | LCZ696(Sacubitril/Valsartan)
Number analyzed (Participants) | 794
Pearson's Correlation Coefficient
  Subjects with new onset HF and/or RAAS naïve: number analyzed (Participants) | 90
  Subjects with new onset HF and/or RAAS naïve | 0.285 [0.083 to 0.465]
  Subjects with HFrEF and "low" NT-proBNP: number analyzed (Participants) | 254
  Subjects with HFrEF and "low" NT-proBNP | 0.201 [0.080 to 0.316]
  Subjects not receiving target dose: number analyzed (Participants) | 204
  Subjects not receiving target dose | 0.165 [0.028 to 0.295]
Statistical Analysis 1: Comparison: LCZ696(Sacubitril/Valsartan); Subjects with new onset HF and/or RAAS naïve; Test type: Other — Pearson's Correlation; p = 0.0060, t-test, 2 sided
Statistical Analysis 2: Comparison: LCZ696(Sacubitril/Valsartan); Subjects with HFrEF and "low" NT-proBNP; Test type: Other — Pearson's Correlation; p = 0.0012, t-test, 2 sided
Statistical Analysis 3: Comparison: LCZ696(Sacubitril/Valsartan); Subjects not receiving target dose; Test type: Other — Pearson's Correlation; p = 0.0181, t-test, 2 sided

8. Secondary Outcome: Change From Baseline in Concentration of N-terminal Pro-brain Natriuretic Peptide (NT-proBNP) and Change in Left Ventricular End Diastolic Volume Index (LVEDVi) by Selected Groups of Interest at Month 6
Description: Pearson's correlation coefficient to examine the association between change in log-transformed NT-proBNP and LVEDVi from baseline to 6 months overall in subgroups of interest, these subgroups are:
  1. Subjects with HFrEF and "low" NT-proBNP (<600 if not hospitalized or <400 if hospitalized) or "low" BNP (<150 if not hospitalized, <100 if hospitalized) at baseline.
  2. Subjects with new onset HF and/or RAAS naïve.
  3. Subjects who are not receiving the target sacubitril/valsartan dose.
Time Frame: Baseline, Month 6
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Pearson's Correlation Coefficient
Arm/Group | LCZ696(Sacubitril/Valsartan)
Number analyzed (Participants) | 794
Pearson's Correlation Coefficient
  Subjects with new onset HF and/or RAAS naïve: number analyzed (Participants) | 90
  Subjects with new onset HF and/or RAAS naïve | 0.122 [-0.087 to 0.321]
  Subjects with HFrEF and "low" NT-proBNP: number analyzed (Participants) | 254
  Subjects with HFrEF and "low" NT-proBNP | 0.123 [0.000 to 0.243]
  Subjects not receiving target dose: number analyzed (Participants) | 204
  Subjects not receiving target dose | 0.078 [-0.060 to 0.213]
Statistical Analysis 1: Comparison: LCZ696(Sacubitril/Valsartan); Subjects with new onset HF and/or RAAS naïve; Test type: Other — Pearson's Correlation; p = 0.2498, t-test, 2 sided
Statistical Analysis 2: Comparison: LCZ696(Sacubitril/Valsartan); Subjects with HFrEF and "low" NT-proBNP; Test type: Other — Pearson's Correlation; p = 0.0495, t-test, 2 sided
Statistical Analysis 3: Comparison: LCZ696(Sacubitril/Valsartan); Subjects not receiving target dose; Test type: Other — Pearson's Correlation; p = 0.2685, t-test, 2 sided

9. Secondary Outcome: Change From Baseline in Concentration of N-terminal Pro-brain Natriuretic Peptide (NT-proBNP) and Change in Left Ventricular Ejection Fraction (LVEF) by Selected Groups of Interest at Month 6
Description: Pearson's correlation coefficient to examine the association between change in log-transformed NT-proBNP and LVEF from baseline to 6 months overall in subgroups of interest, these subgroups are:
  1. Subjects with HFrEF and "low" NT-proBNP (<600 if not hospitalized or <400 if hospitalized) or "low" BNP (<150 if not hospitalized, <100 if hospitalized) at baseline.
  2. Subjects with new onset HF and/or RAAS naïve.
  3. Subjects who are not receiving the target sacubitril/valsartan dose.
Time Frame: Baseline, Month 6
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Pearson's Correlation Coefficient
Arm/Group | LCZ696(Sacubitril/Valsartan)
Number analyzed (Participants) | 794
Pearson's Correlation Coefficient
  Subjects with new onset HF and/or RAAS naïve: number analyzed (Participants) | 90
  Subjects with new onset HF and/or RAAS naïve | -0.308 [-0.484 to -0.107]
  Subjects with HFrEF and "low" NT-proBNP: number analyzed (Participants) | 255
  Subjects with HFrEF and "low" NT-proBNP | -0.202 [-0.317 to -0.081]
  Subjects not receiving target dose: number analyzed (Participants) | 205
  Subjects not receiving target dose | -0.224 [-0.351 to -0.090]
Statistical Analysis 1: Comparison: LCZ696(Sacubitril/Valsartan); Subjects with new onset HF and/or RAAS naïve; Test type: Other — Pearson's Correlation; p = 0.0029, t-test, 2 sided
Statistical Analysis 2: Comparison: LCZ696(Sacubitril/Valsartan); Subjects with HFrEF and "low" NT-proBNP; Test type: Other — Pearson's Correlation; p = 0.0011, t-test, 2 sided
Statistical Analysis 3: Comparison: LCZ696(Sacubitril/Valsartan); Subjects not receiving target dose; Test type: Other — Pearson's Correlation; p = 0.0012, t-test, 2 sided

10. Secondary Outcome: Mean Change in the Kansas City Cardiomyopathy Questionnaire (KCCQ-23) Clinical Summary Score From Baseline to Month 12
Description: The KCCQ-23 is a self-administered questionnaire and requires, on average, 4-6 minutes to complete. It contains 23 items, covering physical function, clinical symptoms, social function, self-efficacy and knowledge, and Quality of Life (QoL). A change of 5 points on the scale scores, either as a group mean difference or an intra-individual change appears to be clinically significant, based on comparisons of changes in the scale scores to clinical indicators and subject global reports of change. The analysis will be done for groups of subjects with N-terminal pro-brain natriuretic peptide<1000 pg/mL and N-Terminal pro-brain natriuretic peptide>=1000 pg/mL at Month 12.
Time Frame: Baseline, month 12
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | LCZ696(Sacubitril/Valsartan)
Number analyzed (Participants) | 794
Points on a scale | 10.39 (19.39)
Statistical Analysis 1: Comparison: LCZ696(Sacubitril/Valsartan); Test type: Other; p < .0001, ANCOVA; Least Squared Mean = 9.32, 95% CI 2-sided [7.94 to 10.69]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment, plus 30 days post treatment, up to maximum duration of approximately 12 months
Description: Any sign or symptom that occurs during the study treatment plus the 30 days post treatment.
Groups:
- LCZ696 (Sacubitril/Valsartan): Subjects received sacubitril/valsartan (LCZ696) on Day 1. The initial dose was determined by the investigator and per the approved indication described in the United States prescribing information/package insert (USPI). The three doses available were: 24/26 mg (Dose Level 1), 49/51mg (Dose Level 2) and 97/103mg (Dose Level 3).
  Titration of the dosage were performed per USPI at 2 to 4 week intervals as clinically tolerated until maximal tolerated or target dosage was achieved. Target dosage was sacubitril/valsartan 97/103 mg twice daily
Arm/Group | LCZ696 (Sacubitril/Valsartan)
All-Cause Mortality (participants affected / at risk) | 30/794
Serious Adverse Events (participants affected / at risk) | 240/794
Other Adverse Events (participants affected / at risk) | 384/794
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LCZ696 (Sacubitril/Valsartan) (N=794)
Anaemia (Blood and lymphatic system disorders) | 5
Coagulopathy (Blood and lymphatic system disorders) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2
Leukocytosis (Blood and lymphatic system disorders) | 1
Acute left ventricular failure (Cardiac disorders) | 3
Acute myocardial infarction (Cardiac disorders) | 7
Angina pectoris (Cardiac disorders) | 8
Atrial fibrillation (Cardiac disorders) | 8
Atrial flutter (Cardiac disorders) | 2
Atrial thrombosis (Cardiac disorders) | 1
Atrioventricular block complete (Cardiac disorders) | 1
Atrioventricular block second degree (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 4
Cardiac failure (Cardiac disorders) | 14
Cardiac failure acute (Cardiac disorders) | 6
Cardiac failure congestive (Cardiac disorders) | 60
Cardiac perforation (Cardiac disorders) | 1
Cardiac ventricular thrombosis (Cardiac disorders) | 3
Cardiogenic shock (Cardiac disorders) | 2
Cardiomyopathy (Cardiac disorders) | 6
Cardiorenal syndrome (Cardiac disorders) | 3
Ischaemic cardiomyopathy (Cardiac disorders) | 3
Left ventricular failure (Cardiac disorders) | 14
Mitral valve incompetence (Cardiac disorders) | 2
Myocardial infarction (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 2
Pericardial effusion (Cardiac disorders) | 1
Pericarditis (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 2
Supraventricular tachycardia (Cardiac disorders) | 5
Ventricular arrhythmia (Cardiac disorders) | 1
Ventricular extrasystoles (Cardiac disorders) | 1
Ventricular fibrillation (Cardiac disorders) | 8
Ventricular tachycardia (Cardiac disorders) | 12
Vertigo (Ear and labyrinth disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 5
Ascites (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 5
Dysphagia (Gastrointestinal disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 5
Gastrointestinal necrosis (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Melaena (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 3
Peptic ulcer (Gastrointestinal disorders) | 1
Retroperitoneal mass (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 3
Spigelian hernia (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Asthenia (General disorders) | 2
Chest pain (General disorders) | 1
Death (General disorders) | 2
Fatigue (General disorders) | 2
Hernia (General disorders) | 1
Medical device site haematoma (General disorders) | 1
Multiple organ dysfunction syndrome (General disorders) | 1
Non-cardiac chest pain (General disorders) | 13
Oedema peripheral (General disorders) | 2
Pain (General disorders) | 1
Peripheral swelling (General disorders) | 1
Physical deconditioning (General disorders) | 1
Pyrexia (General disorders) | 2
Systemic inflammatory response syndrome (General disorders) | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1
Hepatic steatosis (Hepatobiliary disorders) | 1
Hepatitis toxic (Hepatobiliary disorders) | 1
Abscess oral (Infections and infestations) | 1
Arthritis bacterial (Infections and infestations) | 1
Atypical pneumonia (Infections and infestations) | 1
Bacterial sepsis (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 2
Bronchitis viral (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 4
Clostridium difficile colitis (Infections and infestations) | 1
Corona virus infection (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Hepatitis C (Infections and infestations) | 1
Influenza (Infections and infestations) | 3
Localised infection (Infections and infestations) | 3
Osteomyelitis (Infections and infestations) | 6
Periorbital cellulitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 20
Pneumonia bacterial (Infections and infestations) | 1
Pneumonia viral (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 2
Respiratory syncytial virus infection (Infections and infestations) | 1
Respiratory tract infection viral (Infections and infestations) | 1
Sepsis (Infections and infestations) | 7
Septic shock (Infections and infestations) | 4
Staphylococcal infection (Infections and infestations) | 2
Staphylococcal sepsis (Infections and infestations) | 1
Streptococcal infection (Infections and infestations) | 1
Streptococcal sepsis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 7
Vascular device infection (Infections and infestations) | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Brain herniation (Injury, poisoning and procedural complications) | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1
Extradural haematoma (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 5
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 2
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Liver function test increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 5
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1
Failure to thrive (Metabolism and nutrition disorders) | 1
Fluid overload (Metabolism and nutrition disorders) | 2
Fluid retention (Metabolism and nutrition disorders) | 1
Gout (Metabolism and nutrition disorders) | 1
Hyperammonaemia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 9
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Fasciitis (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1
Spondylitis (Musculoskeletal and connective tissue disorders) | 1
Vertebral osteophyte (Musculoskeletal and connective tissue disorders) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder transitional cell carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bone cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ataxia (Nervous system disorders) | 1
Carotid artery disease (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 4
Dizziness (Nervous system disorders) | 4
Embolic cerebral infarction (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 3
Haemorrhage intracranial (Nervous system disorders) | 1
Ischaemic cerebral infarction (Nervous system disorders) | 1
Ischaemic stroke (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 1
Lumbosacral radiculopathy (Nervous system disorders) | 1
Metabolic encephalopathy (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 2
Seizure (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 11
Transient ischaemic attack (Nervous system disorders) | 1
Device failure (Product Issues) | 1
Device malfunction (Product Issues) | 2
Alcohol withdrawal syndrome (Psychiatric disorders) | 1
Bipolar disorder (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Drug abuse (Psychiatric disorders) | 2
Mental status changes (Psychiatric disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 23
Chronic kidney disease (Renal and urinary disorders) | 3
End stage renal disease (Renal and urinary disorders) | 3
Haematuria (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 2
Renal failure (Renal and urinary disorders) | 1
Renal injury (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Ovarian cyst (Reproductive system and breast disorders) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 10
Asthma (Respiratory, thoracic and mediastinal disorders) | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 9
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 10
Angioedema (Skin and subcutaneous tissue disorders) | 3
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 3
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1
Resuscitation (Surgical and medical procedures) | 1
Aortic aneurysm (Vascular disorders) | 1
Aortic stenosis (Vascular disorders) | 1
Circulatory collapse (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Haematoma (Vascular disorders) | 1
Hypertensive crisis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 11
Hypovolaemic shock (Vascular disorders) | 1
Labile blood pressure (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Pelvic venous thrombosis (Vascular disorders) | 1
Peripheral artery stenosis (Vascular disorders) | 1
Peripheral ischaemia (Vascular disorders) | 3
Peripheral venous disease (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LCZ696 (Sacubitril/Valsartan) (N=794)
Diarrhoea (Gastrointestinal disorders) | 43
Fatigue (General disorders) | 56
Oedema peripheral (General disorders) | 44
Upper respiratory tract infection (Infections and infestations) | 58
Blood creatinine increased (Investigations) | 41
Hyperkalaemia (Metabolism and nutrition disorders) | 75
Dizziness (Nervous system disorders) | 129
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 46
Hypotension (Vascular disorders) | 132

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-02-27): https://cdn.clinicaltrials.gov/large-docs/83/NCT02887183/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-22): https://cdn.clinicaltrials.gov/large-docs/83/NCT02887183/SAP_001.pdf